CLINICAL TRIAL: NCT05783817
Title: MDMA-Assisted Cognitive Behavioral Therapy (CBT) Compared With Methamphetamine-Assisted CBT in Obsessive-Compulsive Disorder (OCD): A Phase II Study
Brief Title: MDMA-Assisted CBT for OCD (MDMA-CBT4OCD Study)
Acronym: MDMA-CBT4OCD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Carolyn Rodriguez (Other)
Responsible Party: Sponsor-Investigator, Carolyn Rodriguez, Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 66547
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; MDMA; OCD CBT; Cognitive Behavioral Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Methamphetamine; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized with a 1:1 allocation to either MDMA-assisted CBT or methamphetamine-assisted CBT (active control).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MDMA-assisted cognitive behavioral therapy (Experimental): Administration of 80mg MDMA HCl (with a supplemental dose offered 1.5 to 2 hours later of 40 mg MDMA HCl) in combination with cognitive behavioral therapy (CBT).
  Interventions: Drug: 3,4-Methyl enedioxy methamphetamine; Behavioral: Cognitive Behavioral Therapy (CBT)
- Methamphetamine-assisted cognitive behavioral therapy (Active Comparator): Administration of 10mg methamphetamine (with a supplemental dose offered 1.5 to 2 hours later of 5 mg methamphetamine) in combination with cognitive behavioral therapy (CBT).
  Interventions: Drug: Methamphetamine; Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: 3,4-Methyl enedioxy methamphetamine — MDMA (3,4 methylenedioxymethamphetamine) is a synthetic, psychoactive drug that is chemically similar to the stimulant methamphetamine.
  Other Names: MDMA
  Arms: MDMA-assisted cognitive behavioral therapy
Drug: Methamphetamine — Methamphetamine is a stimulant that affects the central nervous system. This is used as a control in the study.
  Other Names: MA
  Arms: Methamphetamine-assisted cognitive behavioral therapy
Behavioral: Cognitive Behavioral Therapy (CBT) — Cognitive Behavioral Therapy with exposure and response prevention performed by therapist team.

SUMMARY:
The study assesses the safety and preliminary effectiveness of MDMA-assisted cognitive behavioral therapy in participants diagnosed with obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) is a chronic and disabling disorder that costs the economy over $2 billion annually and represents a significant public health problem. The proposed projects tests whether 3,4-Methylenedioxymethamphetamine (MDMA) reduces OCD symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Fluent in speaking and reading the predominantly used or recognized language of the study site
3. Able to swallow pills
4. Meet the criteria for OCD diagnosis
5. YBOCS total score of at least 16
6. Not on psychotropic medications 1 month prior to study enrollment
7. Able to tolerate a treatment-free period
8. Able to tolerate study procedures
9. Failed at least 1 prior trial of standard first-line OCD treatment
10. Agree to the following lifestyle modifications: comply with requirements for fasting and refraining from certain medications prior to the Experimental Session, not enroll in any other interventional clinical trials during the duration of the study, and commit to medication dosing, therapy, and study procedures.

Exclusion Criteria:

1. Pregnant or nursing, or able to become pregnant and are not practicing an effective means of birth control
2. Weigh less than 48 kilograms (kgs)
3. Any current problem which, in the opinion of the investigator or study physician, might interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Chnage in the severity of OCD symptoms as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) | Baseline (Visit 1) to End of Intervention (Visit 13), up to 2 weeks
  Change in OCD severity is measured by the YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response is defined as at least a 35% reduction on the YBOCS.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rodriguez, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mitchell JM, Bogenschutz M, Lilienstein A, Harrison C, Kleiman S, Parker-Guilbert K, Ot'alora G M, Garas W, Paleos C, Gorman I, Nicholas C, Mithoefer M, Carlin S, Poulter B, Mithoefer A, Quevedo S, Wells G, Klaire SS, van der Kolk B, Tzarfaty K, Amiaz R, Worthy R, Shannon S, Woolley JD, Marta C, Gelfand Y, Hapke E, Amar S, Wallach Y, Brown R, Hamilton S, Wang JB, Coker A, Matthews R, de Boer A, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted therapy for severe PTSD: a randomized, double-blind, placebo-controlled phase 3 study. Nat Med. 2021 Jun;27(6):1025-1033. doi: 10.1038/s41591-021-01336-3. Epub 2021 May 10. PMID 33972795